CLINICAL TRIAL: NCT00601562
Title: A Single Dose, Two Treatment, Two Period, Two Sequence, Crossover Bioequivalency Study of 300 mg Zidovudine Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of Zidovudine Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZIDO-04
Record Dates: First submitted 2007-09-19; First posted 2008-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
The objective of this study was to assess the bioequivalence of Roxane's zidovudine 300 mg tablet compared to GlaxoSmithKline's Retrovir® 300 mg tablet under fed conditions using a single-dose, randomized, 2-treatment, 2-period, 2-sequence crossover design.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Participation in a clinical trial within 30 days prior to study initiation.
* Positive blood screen for HIV or Hepatitis B and C.
* History of allergic or adverse responses to zidovudine.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2003-06; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two period, Three day washout

CONTACTS AND LOCATIONS:
Overall Officials: Daniel V Freeland, DO, Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States